CLINICAL TRIAL: NCT05161299
Title: CovidSurg-3: Outcomes of Surgery in COVID-19 Infection
Acronym: CovidSurg-3
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: CovidSurg-3
Record Dates: First submitted 2021-12-16; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: SARS-CoV-2 Infection; Surgery
Keywords: SARS-CoV-2; Surgery; Rapid Antigen test
MeSH Terms: conditions — COVID-19 | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Control (normal practice): Patients that underwent surgery (across all specialities), performed by a surgeon in an operating theatre, AND had a positive SARS-CoV-2 PCR swab or rapid antigen test (if PCR swab is not available) within 7 days before or 30 days after surgery. Patients can be included regardless of whether a specific variant is suspected or unknown
  Interventions: Procedure: Surgery (across all specialities)

INTERVENTIONS:
Procedure: Surgery (across all specialities) — Surgery performed by a surgeon in an operating theatre during the patient inclusion period

SUMMARY:
COVID-19 has significant detrimental impacts on surgical systems and patient outcomes. CovidSurg has provided the best available evidence to guide delivery of safe surgery during the pandemic. However, CovidSurg data were collected in 2020 when the wildtype SARS-CoV-2 virus was dominant, and therefore there is a need to for renewed rapid data to guide global practice during Omicron COVID-19 waves.

CovidSurg-3 is an extension to CovidSurg and was initiated in response to the emergence of the Omicron variant.

CovidSurg-3 has two separate components:

* Patient-level component: Collection of outcome data for patients with peri-operative SARS-CoV-2.
* Hospital-level component: Collection of aggregated case-mix data. Hospitals in countries with low community SARS-CoV-2 infection rates can contribute towards this component.

DETAILED DESCRIPTION:
Data collected in 2020 found patients with perioperative SARS-CoV-2 infection to be at increased risk of postoperative mortality (up to 24% at 30-days), pulmonary complications (up to 51% at 30-days), and venous thromboembolism1-5. Perioperative SARS-CoV-2 infection has been associated with increased mortality, morbidity, longer length of stay, and increased health system burdens compared to SARS-CoV-2 negative patients6-8.

During the first COVID-19 wave, over 28 million elective operations worldwide were either cancelled or delayed9. This enabled redistribution of staff and resources to meet COVID-19 demand, but resulted in substantial treatment delays, including for cancer patients10-11. COVID-19 lockdowns were associated with one in seven patients awaiting cancer surgery not being operated, and those patients who were operated experienced delays10.

In 2020 CovidSurg captured outcomes on over 190,000 patients across >2,000 hospitals in 116 countries. This resulted in data-driven guidance for surgical systems during the pandemic, including:

* Guidance regarding the optimal delay prior to surgery following SARS-CoV-2 infection4.
* The establishment of COVID-19-free surgical pathways to reduce nosocomial infection and complication2.
* The non-effectiveness avoidance of preoperative isolation12.
* Optimal preoperative SARS-CoV-2 screening protocols13.
* Potential benefits of preoperative vaccination14.

The Omicron SARS-CoV-2 variant of concern was first reported on 25 November 2021 and has spread globally rapidly15. There is a high-level of evidence indicating Omicron has increased transmissibility and potential to evade immunity16-18. However, there is little robust evidence regarding disease severity associated with Omicron in both vaccinated and unvaccinated patients (including in surgical patients), nor is there data to guide patient risk stratification during Omicron COVID-19 waves18.

COVID-19 has significant detrimental impacts on surgical systems and patient outcomes. CovidSurg has provided the best available evidence to guide delivery of safe surgery during the pandemic. However, CovidSurg data were collected in 2020 when the wildtype SARS-CoV-2 virus was dominant, and therefore there is a need to for renewed rapid data to guide global practice during Omicron COVID-19 waves.

The primary objective is to determine 30-day mortality in patients with peri-operative SARS-CoV-2 infection. This will inform future risk stratification, decision making, and patient consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients that underwent surgery performed by a surgeon in an operating theatre, AND
* They had a positive SARS-CoV-2 PCR swab or rapid antigen test (if PCR swab is not available) within 7 days before or 30 days after surgery. Patients can be included regardless of whether a specific variant is suspected or unknown

Exclusion Criteria:

* They underwent minor procedures
* Their SARS-CoV-2 infection was diagnosed more than 7 days before surgery (regardless of their symptomatic status at the time of surgery) or beyond 30 days after surgery

All consecutive patients fulfilling inclusion criteria across all specialities should be captured.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that underwent a surgical procedure during the patient inclusion period - 13 December 2021 to 28 February 2022 inclusive, regardless of surgical indication (benign surgery, cancer surgery, trauma, obstetric), anaesthetic type (local, regional, general), surgical approach (minimally invasive surgery, open surgery), or whether it is day-case or in-patient surgery
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-12-13 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-03-29 (Estimated)

PRIMARY OUTCOMES:
To determine 30-day mortality in patients with peri-operative SARS-CoV-2 infection | Up to 30 days post-surgery
  Collection of outcome data (up to 30 days post-surgery) for patients with peri-operative SARS-CoV-2

SECONDARY OUTCOMES:
Rates of post-operative pulmonary complication and venous thromboembolism | Up to 30 days post-surgery
  To determine 30-day postoperative pulmonary complication and venous thromboembolism rates in patients with peri-operative SARS-CoV-2 infection
Evaluate implementation of SARS-CoV-2 mitigations and adaptations (vaccination, preoperative testing, COVID-free surgical pathways, patient selection) | Recruitment period (mid Dec 2021 - end Feb 2022)
  Data collected will help inform future risk stratification and decision making
Frequency of peri-operative SARS-CoV-2 infection | 56 days
  To determine the frequency of peri-operative SARS-CoV-2 infection by collecting aggregated case-mix data at a hospital-level over blocks of 7 consecutive days
Frequency of same-day elective surgery cancellations | 56 days
  To determine the frequency of same-day elective surgery cancellations over blocks of 7 consecutive days

CONTACTS AND LOCATIONS:
Overall Officials: Aneel Bhangu, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No